CLINICAL TRIAL: NCT05449002
Title: Testing a Digital Single-session Intervention for Youths on the Waitlist for Psychotherapy
Brief Title: Digital Single Session Intervention for Youth Mental Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Katherine Venturo-Conerly, Principal Investigator, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB22-0101
Record Dates: First submitted 2022-06-30; First posted 2022-07-08 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Depression; Conduct Disorder; Stress
MeSH Terms: conditions — Anxiety Disorders; Depression; Conduct Disorder

STUDY DESIGN:
Intervention Model Description: Participants, 9-17 years old, will be: randomized to a 30-45-minute Qualtrics-based, digital program teaching Practicing the Opposite (PTO, followed by psychotherapy) or to the usual care (i.e., usual waitlist procedures, followed by psychotherapy) control.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Practicing the Opposite (PTO) intervention (Experimental): This 30-45 minutes Qualtrics-based, digital program uses stories, interactive activities, and engaging graphics to teach youths one core principle: by practicing the positive opposite of unhelpful behaviors (e.g., engaging with rather than avoiding feared stimuli), one can, over time, change their mood, thoughts, and actions. The intervention is comprised of four main sections: 1) An introduction to PTO; (2) Testimonials from young people who have been helped by PTO; (3) Learning how to Practice the Opposite through online activities. (4) Planning how to continue to Practice the Opposite in the participant's life. Of note, after being removed from the waitlist at the clinic and contacted to begin treatment, participants will still receive treatment as usual from the clinic.
  Interventions: Behavioral: Practicing the Opposite (PTO)
- Usual waitlist control group (Other): Usual waitlist procedures involve watchful waiting for a therapist to become available, sometimes complemented by periodic check-ins from the family with clinic administrators. After being removed from the waitlist and contacted to begin treatment, participants in both study conditions will receive treatment as usual in the clinic.
  Interventions: Other: Usual Clinical Care

INTERVENTIONS:
Behavioral: Practicing the Opposite (PTO) — This 30-45-minute digital program is designed to help youths on the waitlist feel better prior to treatment and may also improve their treatment engagement and outcomes.
  Arms: Practicing the Opposite (PTO) intervention
Other: Usual Clinical Care — Usual care provided by participating youth mental health clinics in the United States.
  Arms: Usual waitlist control group

SUMMARY:
The aim of this study is to test the effectiveness of a single-session, digital intervention teaching the principle of practicing the opposite, when administered to youths on the waitlist for psychotherapy, with usual waitlist procedures as a control condition.

DETAILED DESCRIPTION:
There is a massive unmet need for youth mental health care in America; only ¼ of youth in need receive services. The problem has been underscored and exacerbated by the pandemic. The need for child and adolescent mental health care, particularly for depression and anxiety, has surged while clinician availability and clinic funding have shrunk. One result is that clinic waitlists, always lengthy, have stretched, with youths and families who seek care waiting for up to 12 months for a first appointment, and many giving up and dropping out before the much-delayed appointment. There is a clear need-in both pandemic and normal times-for efficient mental health support that can be provided when need is acute, to sustain young people through periods of delayed access, and to reduce burden for professionals. Fortunately, recent evidence shows the surprising potential of brief, low-cost, digital interventions that could go a long way toward bridging the need-to-access gap. Single-session interventions have substantial effects, in some cases rivaling effects of full-length in-person psychotherapy. Remote therapies for youth mental health problems are beneficial on average and approximately as beneficial as in-person psychotherapy.

The current trial will test a brief (one 30-45-minute session), online, interactive mental health and behavior change intervention for adolescents (9-17 years old), who have been placed the waitlist for outpatient treatment at participating mental health clinics in the United States. Previous RCTs show beneficial effects of the principle of Practicing the Opposite (PTO) on youth mental health when using the therapeutic elements present in PTO (e.g., exposure, to overcome anxiety; behavioral activation, to overcome depression). The single-session PTO intervention uses stories, interactive activities, and engaging graphics to teach youths a key principle: by practicing the positive opposite of unhelpful behaviors, one can, over time, change their emotions thoughts, and actions.

ELIGIBILITY:
Inclusion Criteria:

* Youth/family has contacted a participating outpatient clinic to seek mental health care, and is placed on the waitlist.
* Youth is between the ages of 9-17 years (inclusive) at the time of study enrollment.
* Youth and at least one guardian consent to the youth's participation in study.
* Youth reads English well enough to effectively complete the digital programs (defined as taking classes in English, as opposed to ESL classes).
* Youth has access to a digital device.

Exclusion Criteria:

* Youth is non-English speaking, as the program is only available in English.
* Youth does not have access to a digital device.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 226 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Behavior and Feelings Survey (Youth and Parent Versions) | Trajectory of change in scores compared across intervention and control groups from baseline, through post-intervention, 2-week, and monthly follow-up until completion of clinic treatment or 1 year, whichever comes first.
  Assesses the child's thoughts and feelings over the past week using both youth and parent report. Both the youth and parent report surveys include 12 items each scored from 04, with higher scores indicating more severe symptoms. Consists of an internalizing and externalizing subscale, the trajectories of which will be analyzed separately and compared between the intervention and control group. Note that timing described below may be adjusted if response or feedback suggests excessive measurement burden.
Generalized Anxiety Disorder 7-item scale (GAD-7) | Trajectory of change in scores compared across intervention and control groups from baseline, through post-intervention, 2-week, and monthly follow-up until completion of clinic treatment or 1 year, whichever comes first.
  Assesses via a 7-item youth self-report questionnaire (in which scores range from 0-21, and higher scores indicate more severe symptoms) the youth's experience of anxiety symptoms. Trajectory of change on this measure will be compared between the intervention and control group. Note that timing described below may be adjusted if response or feedback suggests excessive measurement burden.
Patient Health Questionnaire 8-item scale (PHQ-8) | Trajectory of change in scores compared across intervention and control groups from baseline, through post-intervention, 2-week, and monthly follow-up until completion of clinic treatment or 1 year, whichever comes first.
  Assesses via an 8-item youth self-report questionnaire (in which scores range from 0-24, and higher scores indicate more severe symptoms) the youth's experience of anxiety symptoms. Trajectory of change on this measure will be compared between the intervention and control group. Note that timing described below may be adjusted if response or feedback suggests excessive measurement burden.
Revised Children's Anxiety and Depression Scale (RCADS) Parent Version (Short Form) | Trajectory of change in scores compared across intervention and control groups from baseline, through post-intervention, 2-week, and monthly follow-up until completion of clinic treatment or 1 year, whichever comes first.
  Trajectory of change on this 24-item parent-report measure of anxiety and depression (in which scores range from 0-72 and higher scores indicate more severe symptoms) will be compared between the intervention and control group. Trajectories of change on the subscales within this measure (broad anxiety and depression) may also be analyzed similarly. Note that timing described below may be adjusted if response or feedback suggests excessive measurement burden.

SECONDARY OUTCOMES:
Ecological Momentary Assessment (EMA) Survey | Scores on each item will be compared across 1 week before the PTO intervention and 2-weeks after. The association between change in behaviors and change in affect across these time ranges will be assessed.
  Consisting of a modified Positive and Negative Affect Scale (PANAS) and a modified Coping Questionnaire, this 8-item measure is administered 3 times daily via an EMA mobile application called Metricwire. It assesses affect and behaviors via youth self-report.
State Hope Scale | Trajectory of change in scores compared across intervention and control groups from baseline, through post-intervention, 2-week, and 1-month follow-up.
  Assesses the child's current level of hope using a six-item self-report scale, in which each item is scored from 1 to 8, with higher scores indicating greater hope. Trajectory of change on this measure will be compared between the intervention and control group. Note that timing described below may be adjusted if response or feedback suggests excessive measurement burden.
Perceived Control Scale for Children | Trajectory of change in scores compared across intervention and control groups from baseline, through post-intervention, 2-week, and 1-month follow-up.
  Assesses via a 24-item self-report scale the youth's beliefs about their ability to control and change their environment. Total scores range from 0-72, with higher scores indicating greater perceived control. Trajectory of change on this measure will be compared between the intervention and control group. Note that timing described below may be adjusted if response or feedback suggests excessive measurement burden.
Secondary Control Scale for Children | Trajectory of change in scores compared across intervention and control groups from baseline, through post-intervention, 2-week, and 1-month follow-up.
  Assesses via a 20-item self-report scale the youth's beliefs about their ability to control and change their emotions and thoughts. Total scores range from 0-60, with higher scores indicating greater secondary control. Trajectory of change on this measure will be compared between the intervention and control group. Note that timing described below may be adjusted if response or feedback suggests excessive measurement burden.
Clinic Record Data | Through study completion, an anticipated average of 6-months
  For those participants who authorize investigator access to their clinic record data, the investigators will also compare rates of accessing and completing clinic treatment, as well as attendance at sessions, between the intervention and control groups.

OTHER OUTCOMES:
Feedback Questionnaire | immediately post-intervention
  Elicits feedback from the youth about the digital practicing the opposite program.
Demographic Questionnaire | pre-intervention
  Asks caregiver and youth for basic youth and family demographic information.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Venturo-Conerly, A.B., Principal Investigator — Harvard University
Locations (5):
- United States (5):
  - Riley Child Psychiatry and Behavioral Sciences Clinic, Indianapolis, Indiana
  - Boston Child Study Center, Boston, Massachusetts
  - The Baker Center for Children and Families, Boston, Massachusetts
  - The Concord Center, Concord, Massachusetts
  - Riverside Community Care, Dedham, Massachusetts